CLINICAL TRIAL: NCT05294549
Title: Implementation of Caring Contacts Using Patient Feedback to Reduce Suicidal Ideation Following Psychiatric Hospitalization
Brief Title: Implementation of Caring Contacts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Rosalie Steinberg, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5262
Record Dates: First submitted 2022-03-07; First posted 2022-03-24 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Psychiatric Hospitalization
Keywords: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caring Contact (Experimental)
  Interventions: Other: Caring Contact

INTERVENTIONS:
Other: Caring Contact — The Caring Contact intervention is an email with messages of hope, support and resource information sent to patients post-discharge from psychiatric hospitalization.

SUMMARY:
This quality improvement (QI) project will adapt and improve an evidence-based suicide-prevention initiative for Sunnybrook patients at high risk of suicide following psychiatric inpatient discharge, targeting one of Sunnybrook's QI Plan goals of reducing suicide at Sunnybrook. Caring Contacts, brief communications of hope, support and information sent to patients post-discharge, are a simple and low-cost intervention with proven effectiveness in reducing suicide attempts, suicidal ideation, and loneliness, while increasing hopefulness and feelings of connection to the health care system. Pilot data provides some initial, promising evidence however additional patient input is required to improve the acceptability and effectiveness of the intervention to reduce suicide-related outcomes. Feedback from patients and peer advisors will guide iterative improvements with the ultimate goal of implementing an improved version of Caring Contacts as a standard clinical practice for all patients discharged from the Sunnybrook Adult Inpatient Psychiatry Unit.

For phase one of this QI project, participants will be patients from the Sunnybrook Inpatient Psychiatry Unit with suicidality and community members with lived experience of psychiatric hospitalization and suicidality. Investigators will conduct focus groups on the inpatient unit of 8-12 inpatient participants to gather feedback about the current Caring Contact intervention. For community members virtual focus groups will be conducted. For phase two, participants will be patients from the Sunnybrook Inpatient Psychiatry Unit with suicidality. The updated intervention will be sent to 8-12 participants. Then investigators will host virtual focus groups to gather feedback from these participants about the intervention. For phase three, participants will be patients from the Sunnybrook Inpatient Psychiatry Unit with suicidality. Investigators will send the revised intervention to 30-40 participants. Participants will complete symptom and feedback questionnaires when they receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Age 18 or above
3. Ability to read and understand English
4. Have an email address
5. The ability to understand and comply with the requirements of the project and capable of providing informed consent

For inclusion in the outpatient focus groups participants must additionally have previous lived experience of psychiatric hospitalization with suicidal ideation or behaviour.

For inclusion in the inpatient focus groups during phase one and for inclusion in the second and third phases of the project, participants must additionally 1) be an inpatient on the Sunnybrook Adult Inpatient Psychiatry Unit at the time of recruitment and 2) they must have been admitted to the unit with suicidal ideation or behaviour as determined by their C-SSRS score at admission.

Exclusion Criteria:

* A primary diagnosis of a Major Neurocognitive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Feedback questionnaire | Through study completion about 1 year
  Feedback questionnaire responses using Likert scales will be quantified and compared as a measure of acceptability of the intervention.
Focus group responses | Through first 3 months of study
  Qualitative thematic analyses will be used to evaluate the focus group transcripts.
Hopkins Symptom Checklist-25 (HSCL-25) | Baseline, up to 14 days post-discharge
  The HSCL-25 is a widely used self-report questionnaire using a Likert scale to measure mood symptoms. The HSCL-25 has an item for suicidal ideation. Total change scores and suicidal ideation change scores will be used to assess the effectiveness of intervention.
  Minimum total score is 25, maximum is 100. A higher score equals a worse outcome.
The Entrapment Scale | Baseline, up to 14 days post-discharge
  The Entrapment scale is a 16 item scale used to identify feelings of entrapment, which is a driver for suicidal behaviour. Total change scores will be used to assess the effectiveness of the intervention. Minimum total score is 0, maximum is 80. A higher score equals a worse outcome.
Beck Scale for Suicidal Ideation (BSI) | Baseline, up to 14 days post-discharge
  The BSI is a self-report questionnaire with 21 items used to detect and measuring the current intensity of an individual's attitudes, behaviors, and plans to commit suicide during the past week. Total change scores will be used to assess the effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada